CLINICAL TRIAL: NCT04472000
Title: Can Vitamin C Reduce the Risk of Postoperative Shoulder Stiffness? A Multi-center, Double-blinded, Randomized and Placebo-controlled Study
Brief Title: Can Vitamin C Reduce the Risk of Postoperative Shoulder Stiffness?
Acronym: VitC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study had to be stopped due to difficulties in recruiting patients.
Sponsor: Lindenhofgruppe AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-00605
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Shoulder Stiffness
Keywords: Vitamin C; pain; mobility; rotation; glenohumeral joint
MeSH Terms: conditions — Pain | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to the two treatment arms, vitamin C or placebo, in a 1:1 ratio. The randomisation will be stratified by type of surgery performed. Allocation will be concealed using sequentially coded drug packs that are otherwise identical. Drug packs will be coded as 01-01 to 01-50 for stratum 1, 02-01 to 02-50 for stratum 2, 03-01 to 03-50 for stratum 3, and 04-01 to 04-50 for stratum 4.
  The 4 strata differ in the type of operation performed:
  1. Rotator cuff surgery with resection of the acromioclavicular joint
  2. Rotator cuff surgery without resection of the acromioclavicular joint
  3. Shoulder arthroscopy with resection of the acromioclavicular joint
  4. Shoulder arthroscopy without resection of the acromioclavicular joint Vitamin C will be administered orally at 1000 mg/day (500 mg b.i.d.) for 50 days post surgery.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All study participants and trial personnel but the persons generating the randomization list and preparing the blinded drug packs at the Inselapotheke and Spitalapotheke Lindenhof will be blinded to the assigned treatment. Blinding will be upheld until all analyses are completed. Vitamin C and placebo will be provided in identical looking capsules in drug packs, which will also look identical except for the consecutive code number which is unique on each pack.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin C (Experimental): Patients who are assigned to the experimental treatment group will be given extended release capsules with 500 mg of ascorbic acid orally two times daily, packed in PET/PP-bottles identical as used for the licenced product.
  Interventions: Drug: Vitamin C
- Placebo (Placebo Comparator): The control intervention of this study consists of treatment with no active substance (placebo) but in the same schedule as the experimental treatment (verum).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin C — Study participants in the verum group receive one capsule of Burgerstein Vitamin C retard 500mg b.i.d. with treatment starting in the evening on the day of the operation for a total of 50 days.
  Arms: Vitamin C
Drug: Placebo — The placebo group receives one placebo capsule b.i.d. with treatment starting in the evening on the day of the operation for a total of 50 days.
  Arms: Placebo

SUMMARY:
Postoperative shoulder stiffness is a common complication after shoulder surgery (incidence 10-15%). The symptoms consist primarily in a painful impairment of the mobility of the glenohumeral joint, usually after initially good course. Cause and origin are not clear.

Vitamin C is known as an inactivator of free radicals and plays a key role in building collagen tissue. Vitamin C thus has a modulating role in inflammatory reactions. Injured and ill people have been shown to have significantly increased vitamin C needs, which underlines this role. Evidence was also found that vitamin C has a positive influence on similar diseases such as the complex regional pain syndrome (CRPS, Morbus Sudeck) on the wrist and postoperative arthrofibrosis on the knee joint.

The Investigators want to investigate whether vitamin C intake can positively influence the incidence and / or severity of postoperative shoulder stiffness after shoulder surgery.

The primary objective of this study is to investigate the effect of vitamin C on the external rotational ability of the operated shoulder in the glenohumeral joint compared to the opposite side at 12 weeks post surgery.

Secondary objectives of this study are to investigate other shoulder mobility tests, patient-reported outcomes (level of pain, ability/return to work, smoking habits), patient-reported questionnaires (Constant Score, Oxford shoulder score, DASH score) and the incidence of a frozen shoulder at 6, 12, 26, and 52 weeks post surgery.

Total duration of study: 2.5 years.

DETAILED DESCRIPTION:
Participants will be randomly allocated to the two treatment arms, vitamin C or placebo, in a 1:1 ratio Study participants in the verum group receive one capsule of Burgerstein Vitamin C retard 500mg b.i.d. with treatment starting in the evening on the day of the operation for a total of 50 days.

The placebo group receives one placebo capsule b.i.d. with treatment starting in the evening on the day of the operation for a total of 50 days. Vitamin C will be administered orally. Burgerstein Vitamin C Retard Capsules 500 mg (Pharmacode: 6739189) will be used for this study. Active substance: Ascorbic acid (Vitamin C, E 300).

Since a known drug should be tested for a new indication, the exclusion of a bias by a placebo effect, the administration of a placebo to the control group is necessary. To exclude a detection bias and a performance bias, the study is performed double-blind. A randomization protects against a selection bias.

The determination of the sample size is based on the following considerations. The primary endpoint is not expected to be normally distributed. Therefore the sample size determination is based on a Mann-Whitney test for the comparison of the two groups (placebo and treatment) assuming a logistic distribution. Based on a few data of comparable measurements the Investigators think that the standard deviation of the primary endpoint is 10(=SD) in each group. The treatment effect is expected to be Delta=10, a medically reasonable effect.

To achieve a power of at least 80% for the 4 tested comparisons in the final analysis of the primary endpoint, a minimal sample size of 42 in each of the 4 patient groups (strata) is required. In expectation of a drop-out rate of 20%, the target sample size will be 50 patients in each stratum and 200 patients in total, with 100 in the placebo group and 100 in the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* 18 years or older at the time of informed consent signature
* Complication-free rotator cuff* or shoulder arthroscopy** with or without resection of the acromioclavicular joint at the orthopedics Sonnenhof. The rotator cuff operations are basically open or in mini-open technique, usually with additional tenotomy / tenodesis of the long biceps tendon.

  * rotator cuff surgery can include tenotomy/tenodesis of long biceps tendon, intra-articular debridement with or without resection of the coracoacromial ligament and/or acromioplasty, biopsies, diagnostic arthroscopy

  ** Arthroscopic procedures include subacromial debridement (including partial resection of the coracoacromial ligament & acromioplasty), diagnostic arthroscopy, tenotomy of the long biceps tendon, intra-articular debridement, resection of calcium depots for treatment of tendinitis calcarea, biopsies, stabilizations (only without postoperative immobilization)
* Sufficient knowledge of German to understand the patient information and informed consent, follow instructions by study personnel, and complete patient questionnaires & diary

Exclusion Criteria:

* Contraindications to ascorbic acid or one of the excipients, e.g. known hypersensitivity or allergy to the investigational product
* Planned single or multiple intake of vitamin supplements during the study period, which results in an additional daily intake of > 50 mg ascorbic acid
* Known pregnancy or breast feeding
* Known or suspected non-compliance, for example drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to psychological disorders, dementia, etc.
* Participation in another interventional study within the 30 days preceding and during the present study
* Previous enrollment into the current study
* Enrollment of the investigator, his / her family members, employees and other dependent persons
* Current or previous frozen shoulder (no matter on which side)
* Pre-surgery on the affected shoulder joint (preoperative procedures include all procedures examined in this study, including all other procedures involving the glenohumeral joint and / or acromioclavicular joint. In addition, all interventions, which as a result, negatively influence the mobility of the shoulder with great likelihood up to the current time)
* Known current unstable medical problem on the not-affected shoulder joint according to the judgment of the investigator
* Taking a cortisone preparation or an immunomodulatory drug (for example methotrexate or similar)
* Alcoholism (defined as intake of more than 12g (women) or 24g (men) alcohol per day)
* Regular hemodialysis
* Known diabetes mellitus
* Known Addison's disease
* Known not correctly adjusted thyroid metabolism
* Known Parkinson's disease and similar CNS disorders (Diffuse Lewy Body Disease, Corticobasal Degeneration, Multisystem Atrophy, Progressive Supranuclear Paralysis, Essential Tumor, Huntington's Disease, Multiple Sclerosis)
* Known diseases / injuries of the peripheral nerves (Isaac's Syndrome, Stiff-Person Syndrome, Guillain-Barré Syndrome, Chronic Inflammatory Demyelinating Polyneuropathy, Hereditary Neuropathies, Amyotrophic Lateral Sclerosis, Hereditary Motor Neuropathies Prone to Pressure Paralysis, Motor Neurone Diseases, Myasthenia Gravis, Spinal Muscular Atrophies, Thoracic Outlet Syndromes)
* Known infection in the shoulder joint to be operated
* Known Hyperlipidemia
* Known Uremia
* Known Thalassemia
* Known iron storage diseases
* Known Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Planned further operation of any kind within the next 50 days after shoulder surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2024-04-21 (Actual)

PRIMARY OUTCOMES:
Difference between the external glenohumeral joint rotations of the operated shoulder and the opposite shoulder | 12 weeks post surgery
  The primary endpoint of this study is the difference between the external glenohumeral joint rotations of the operated shoulder and the opposite shoulder ("Delta ∆").
  The external glenohumeral joint rotation was chosen as primary measure for shoulder performance because this is the component of movement in the shoulder joint, which is the first and most severely impaired in postoperative shoulder stiffness and which normalizes as the last after the symptomatology subsides.
  Delta ∆ was chosen as an outcome measure, since the standard deviation of the external rotation capability in the population is very high. The external glenohumeral joint rotation of both shoulders is measured using a smartphone with the App "GetMyROM".

SECONDARY OUTCOMES:
Delta ∆ of the external glenohumeral joint rotation | after 6, 26, and 52 weeks post surgery
  The external glenohumeral joint rotation of both shoulders is measured using a smartphone with the App "GetMyROM"
Delta ∆ of abduction | after 6, 26, and 52 weeks post surgery
  - Abduction will be assessed using the GetMyROM-App. Abduction will be done passively with the glenohumeral joint fixed.
Delta ∆ of internal rotation | after 6, 26, and 52 weeks post surgery
  -Internal rotation will be assessed using typical landmarks in clinical practice (Trochanter major, Gluteus maximus/Buttocks, Belt, lumbar spine, thoracolumbar junction, breast spine, interscapular)
Delta ∆ of flexion | after 6, 26, and 52 weeks post surgery
  -Flexion will be assessed using the GetMyROM-App. Flexion will be done passively with the glenohumeral joint fixed.
Level of pain | daily during the first 50 days post surgery, and at 12, 26, and 52 weeks post surgery as a criterion for the occurrence of postoperative frozen shoulder
  Secondary endpoints include the Level of pain of the operated shoulder preoperatively and level of pain (at rest and in motion) will be assessed using the VAS pain scale
Work ability | 6, 26, and 52 weeks post surgery
  Secondary endpoints include work ability (back-to-work ratio) post surgery. The (partial) ability to work is requested.
Oxford shoulder score | preoperatively and after 6, 12, 26, and 52 weeks
  Secondary endpoints include the Oxford shoulder score as a measure of the pain and the utilizability of the shoulder as well as the patient satisfaction. Will be recorded by the patient getting a questionnaire, which he or she fills out in the waiting room before the appointment with the doctor. The practical part of the Constant score is subsequently filled in by the doctor during the clinical follow-up examination.
Constant Score | preoperatively and depending on the procedure after 6 and 12 weeks (strata 3 & 4), and after 26 and 52 weeks (all strata)
  Secondary endpoints include the Constant Score as a measure of everyday utilizability of the shoulder and patient satisfaction. Will be recorded by the patient getting a questionnaire, which he or she fills out in the waiting room before the appointment with the doctor. The practical part of the Constant score is subsequently filled in by the doctor during the clinical follow-up examination. The Force measurement in the Constant score is performed with the following device: IsoForceControl®EVO2 - Dynamometer 10-400N.
DASH score | preoperatively and after 6, 12, 26, and 52 weeks
  Secondary endpoints include the DASH score as a measure of the pain and the utilizability of the shoulder as well as the patient satisfaction. Will be recorded by the patient getting a questionnaire, which he or she fills out in the waiting room before the appointment with the doctor. The practical part of the Constant score is subsequently filled in by the doctor during the clinical follow-up examination.
Smoking habits | end of the study, up to 2.5 years
  Secondary endpoints include the influence of smoking habits on the outcome and possibly on the effect of the study drug. The (current) smoking habits are documented.
Frozen shoulder | end of the study, up to 2.5 years
  Secondary endpoints include the incidence of frozen shoulder. There is no standard definition for frozen shoulder in the literature. The diagnosis is made clinically. The frozen shoulder in this study is defined as a further decrease in external rotation of the glenohumeral joint in the postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Janine Antonov, Dr., Study Chair — Campus SLB, Lindenhof AG
Locations (2):
- Switzerland (2):
  - Spital Aaberg, Aarberg, Canton of Bern
  - Orthopädie Sonnenhof, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho CH, Song KS, Kim BS, Kim DH, Lho YM. Biological Aspect of Pathophysiology for Frozen Shoulder. Biomed Res Int. 2018 May 24;2018:7274517. doi: 10.1155/2018/7274517. eCollection 2018. PMID 29992159
- [Background] Wong CK, Levine WN, Deo K, Kesting RS, Mercer EA, Schram GA, Strang BL. Natural history of frozen shoulder: fact or fiction? A systematic review. Physiotherapy. 2017 Mar;103(1):40-47. doi: 10.1016/j.physio.2016.05.009. Epub 2016 Jun 21. PMID 27641499
- [Background] Kim DH, Kim YS, Kim BS, Sung DH, Song KS, Cho CH. Is frozen shoulder completely resolved at 2 years after the onset of disease? J Orthop Sci. 2020 Mar;25(2):224-228. doi: 10.1016/j.jos.2019.03.011. Epub 2019 Apr 2. PMID 30952550
- [Background] Aim F, Klouche S, Frison A, Bauer T, Hardy P. Efficacy of vitamin C in preventing complex regional pain syndrome after wrist fracture: A systematic review and meta-analysis. Orthop Traumatol Surg Res. 2017 May;103(3):465-470. doi: 10.1016/j.otsr.2016.12.021. Epub 2017 Mar 4. PMID 28274883
- [Background] Kim JH, Kim YC, Nahm FS, Lee PB. The Therapeutic Effect of Vitamin C in an Animal Model of Complex Regional Pain Syndrome Produced by Prolonged Hindpaw Ischemia-Reperfusion in Rats. Int J Med Sci. 2017 Jan 15;14(1):97-101. doi: 10.7150/ijms.17681. eCollection 2017. PMID 28138314
- [Background] Chen S, Roffey DM, Dion CA, Arab A, Wai EK. Effect of Perioperative Vitamin C Supplementation on Postoperative Pain and the Incidence of Chronic Regional Pain Syndrome: A Systematic Review and Meta-Analysis. Clin J Pain. 2016 Feb;32(2):179-85. doi: 10.1097/AJP.0000000000000218. PMID 25654537
- [Background] Fukushima R, Yamazaki E. Vitamin C requirement in surgical patients. Curr Opin Clin Nutr Metab Care. 2010 Nov;13(6):669-76. doi: 10.1097/MCO.0b013e32833e05bc. PMID 20689415
- [Background] Behrend H, Lengnick H, Zdravkovic V, Ladurner A, Rudin D, Erschbamer M, Joerger M, Kuster M. Vitamin C demand is increased after total knee arthroplasty: a double-blind placebo-controlled-randomized study. Knee Surg Sports Traumatol Arthrosc. 2019 Apr;27(4):1182-1188. doi: 10.1007/s00167-018-5030-3. Epub 2018 Jun 28. PMID 29955932
- [Background] Giladi AM, Dossett LA, Fleming SB, Abumrad NN, Cotton BA. High-dose antioxidant administration is associated with a reduction in post-injury complications in critically ill trauma patients. Injury. 2011 Jan;42(1):78-82. doi: 10.1016/j.injury.2010.01.104. Epub 2010 Feb 10. PMID 20149369
- [Background] Rizzo JA, Rowan MP, Driscoll IR, Chung KK, Friedman BC. Vitamin C in Burn Resuscitation. Crit Care Clin. 2016 Oct;32(4):539-46. doi: 10.1016/j.ccc.2016.06.003. Epub 2016 Aug 2. PMID 27600125
- [Background] Kleszczewski T, Modzelewska B, Lisowska A, Buzun L, Kleszczewska E. Levels of vitamin C In the blood plasma patients treated with coronary artery bypass grafting increases significantly after surgery. Biomed Pharmacother. 2017 Jan;85:527-530. doi: 10.1016/j.biopha.2016.11.060. Epub 2016 Nov 24. PMID 27890433
- [Background] Lee GW, Yang HS, Yeom JS, Ahn MW. The Efficacy of Vitamin C on Postoperative Outcomes after Posterior Lumbar Interbody Fusion: A Randomized, Placebo-Controlled Trial. Clin Orthop Surg. 2017 Sep;9(3):317-324. doi: 10.4055/cios.2017.9.3.317. Epub 2017 Aug 4. PMID 28861199
- [Background] Zollinger PE, Tuinebreijer WE, Breederveld RS, Kreis RW. Can vitamin C prevent complex regional pain syndrome in patients with wrist fractures? A randomized, controlled, multicenter dose-response study. J Bone Joint Surg Am. 2007 Jul;89(7):1424-31. doi: 10.2106/JBJS.F.01147. PMID 17606778
- [Background] Zollinger PE, Tuinebreijer WE, Kreis RW, Breederveld RS. Effect of vitamin C on frequency of reflex sympathetic dystrophy in wrist fractures: a randomised trial. Lancet. 1999 Dec 11;354(9195):2025-8. doi: 10.1016/S0140-6736(99)03059-7. PMID 10636366
- [Background] Traxer O, Huet B, Poindexter J, Pak CY, Pearle MS. Effect of ascorbic acid consumption on urinary stone risk factors. J Urol. 2003 Aug;170(2 Pt 1):397-401. doi: 10.1097/01.ju.0000076001.21606.53. PMID 12853784
- [Background] Thomas LD, Elinder CG, Tiselius HG, Wolk A, Akesson A. Ascorbic acid supplements and kidney stone incidence among men: a prospective study. JAMA Intern Med. 2013 Mar 11;173(5):386-8. doi: 10.1001/jamainternmed.2013.2296. No abstract available. PMID 23381591
- [Background] Prier M, Carr AC, Baillie N. No Reported Renal Stones with Intravenous Vitamin C Administration: A Prospective Case Series Study. Antioxidants (Basel). 2018 May 21;7(5):68. doi: 10.3390/antiox7050068. PMID 29883396
- [Background] Mitch WE, Johnson MW, Kirshenbaum JM, Lopez RE. Effect of large oral doses of ascorbic acid on uric acid excretion by normal subjects. Clin Pharmacol Ther. 1981 Mar;29(3):318-21. doi: 10.1038/clpt.1981.42. PMID 7471601
- [Background] Auer BL, Auer D, Rodgers AL. The effect of ascorbic acid ingestion on the biochemical and physicochemical risk factors associated with calcium oxalate kidney stone formation. Clin Chem Lab Med. 1998 Mar;36(3):143-7. doi: 10.1515/CCLM.1998.027. PMID 9589801
- [Background] Levine M, Conry-Cantilena C, Wang Y, Welch RW, Washko PW, Dhariwal KR, Park JB, Lazarev A, Graumlich JF, King J, Cantilena LR. Vitamin C pharmacokinetics in healthy volunteers: evidence for a recommended dietary allowance. Proc Natl Acad Sci U S A. 1996 Apr 16;93(8):3704-9. doi: 10.1073/pnas.93.8.3704. PMID 8623000
- [Background] Padayatty SJ, Levine M. Vitamin C: the known and the unknown and Goldilocks. Oral Dis. 2016 Sep;22(6):463-93. doi: 10.1111/odi.12446. Epub 2016 Apr 14. PMID 26808119
- [Background] Zhang M, Jativa DF. Vitamin C supplementation in the critically ill: A systematic review and meta-analysis. SAGE Open Med. 2018 Oct 19;6:2050312118807615. doi: 10.1177/2050312118807615. eCollection 2018. PMID 30364374
- [Background] Gerster H. No contribution of ascorbic acid to renal calcium oxalate stones. Ann Nutr Metab. 1997;41(5):269-82. doi: 10.1159/000177954. PMID 9429689
- [Background] Zuckerman JD, Rokito A. Frozen shoulder: a consensus definition. J Shoulder Elbow Surg. 2011 Mar;20(2):322-5. doi: 10.1016/j.jse.2010.07.008. Epub 2010 Nov 4. PMID 21051244
- [Background] Mejia-Hernandez K, Chang A, Eardley-Harris N, Jaarsma R, Gill TK, McLean JM. Smartphone applications for the evaluation of pathologic shoulder range of motion and shoulder scores-a comparative study. JSES Open Access. 2018 Mar 13;2(1):109-114. doi: 10.1016/j.jses.2017.10.001. eCollection 2018 Mar. PMID 30675577